CLINICAL TRIAL: NCT01912807
Title: Intravenous Dextrose Versus Ondansetron for Prevention of Postoperative Vomiting in Children: a Randomized Non-inferiority Trial
Brief Title: Postoperative Vomiting in Children - Is Dextrose an Effective Prophylactic Anti-emetic?
Acronym: DEXPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Andrea Vasquez, Clinical Assistant Professor - University of Saskatchewan, Department of Academic Family Medicine, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-163
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Vomiting
Keywords: Postoperative vomiting; Children
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glucose; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dextrose (D5NS) (Experimental): The participants received Dexamethasone (dose 0,15 mg/Kg) as standard antiemetic prophylaxis and Dextrose 5% in 0.9 % Normal Saline (D5NS) was used as a second antiemetic, at an intravenous rate calculated based on their weight and determined for the purpose of the study.
  Interventions: Drug: Dextrose (D5NS)
- Ondansetron (Control) (Active Comparator): The control group received Dexamethasone (dose 0,15 mg/Kg) as standard antiemetic prophylaxis. Ondansetron (dose 0,05 mg/Kg) was used as a second prophylactic antiemetic.
  Interventions: Drug: Ondansetron (Control)

INTERVENTIONS:
Drug: Dextrose (D5NS) — Solution Dextrose 5% in Normal Saline (D5NS) was used as a second antiemetic, at an intravenous maintenace rate (4 cc per Kg for first 10 Kg, 2 cc per Kg for next 10 Kg and 1 cc per Kg for the next Kg of weight) calculated based on the patient's weight
  Other Names: Dextrose 5% in 0,9% Normal Saline
  Arms: Dextrose (D5NS)
Drug: Ondansetron (Control) — Ondansetron was used at a prophylactic dose (0,05 mg per Kg) based on patient's weight.
  Other Names: Zofran
  Arms: Ondansetron (Control)

SUMMARY:
The aim of this study was to investigate the efficacy of intraoperative intravenous dextrose in preventing POV in pediatric population undergoing dental day surgery.

Post-operative vomiting (POV) in children is a frequent complication. Studies using intravenous (IV) fluids containing dextrose in the perioperative period have shown improvement of POV in adults. Similar studies have not been done in children.

Knowing that Intravenous (IV) fluids containing dextrose are safe and commonly used in the paediatric population, this intervention could potentially reduce the amount of rescue antiemetic medications and improve recovery in same-day surgery paediatric patients.

DETAILED DESCRIPTION:
A non-inferiority randomized control trial of healthy children (3-9 years old) undergoing ambulatory dental surgery was conducted to investigate the efficacy of intraoperative IV fluids containing dextrose for antiemetic prophylaxis.

The control group (146 participants) received dexamethasone (0.15 mg/kg IV) and ondansetron (0.05 mg/kg IV); the intervention group (144) received dexamethasone (0.15 mg/kg IV) and intravenous 5% dextrose in 0.9% normal saline (D5NS) as per a weight based maintenance rate.

Patients underwent a general anesthetic maintained with a volatile anesthetic. There was not a standardized protocol for anesthetic induction and maintenance, and all types and doses of anesthetic medications were chosen and administered at the discretion of the anesthesiologist. Intraoperative administration of any other antiemetic medications constituted protocol violation and excluded the patient from analysis. There were no modifications to the planned dental procedure.

Once IV access was established and the patient was intubated, the maintenance study solution was connected and infused throughout the operative period. Additional fluid (Ringer's Lactate) was available to the anesthesiologists to administer as per their preference.

The study drug was administered to the patient by the anesthesiologist at the end of the procedure, when the throat packing was removed and the IV maintenance study solution was stopped. Before emergence from anesthesia, the researcher measured and recorded the patient's blood sugar via a chemstrip (AccuCheck aviva ®). Ringer's Lactate IV fluid, not part of study protocol, was continued in recovery based on the anesthesiologist's preference.

All patients were transferred to the post-anesthetic care unit (PACU) at the end of the procedure. Discharge from the PACU was based on the Post Anesthetic Discharge Scoring System (PADSS) and institutional guidelines. Nursing staff and researchers recorded the presence and incidence of POV in the PACU. Analgesics and antiemetic agents were prescribed by the anesthesiologist during the recovery period and given according to nursing assessment based on institutional guidelines.

Researchers phoned participants 24 hours after discharge to inquire about incidence of emesis and any need to seek medical attention after being discharged from the institution.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 9 Years of age
* Male and Female
* ASA I and II
* Paediatric patients undergoing same-day dental procedures at the Prairieview Surgical Centre.

Exclusion Criteria:

* Age <3 or >9
* Underlying pro-emetic disease
* Positive history of POV in the patient, parent or sibling
* Currently on antiemetic medications
* Parent refusal to sign consent
* History of juvenile diabetes

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vasquez, MD, Principal Investigator — University of Saskatchewan; Jonathan Gamble, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Prairieview Surgical Centre, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Vasquez-Camargo A, Gamble J, Fedoruk KA, Lim HJJ, Mondal PK, Martinez J, Miller GG. Intravenous dextrose versus ondansetron for prevention of postoperative vomiting in children: a randomized non-inferiority trial. Can J Anaesth. 2020 Oct;67(10):1333-1340. doi: 10.1007/s12630-020-01757-7. Epub 2020 Jul 21. PMID 32696227

RESULTS

PARTICIPANT FLOW:
Groups:
- Dextrose (D5NS) - Intervention Group: The participants received Dexamethasone (dose 0,15 mg/Kg) as standard antiemetic prophylaxis and Dextrose 5% in 0.9 % Normal Saline (D5NS) was used as a second antiemetic, at an intravenous rate calculated based on their weight and determined for the purpose of the study.
  Dextrose (D5NS): Solution Dextrose 5% in Normal Saline (D5NS) was used as a second antiemetic, at an intravenous maintenace rate (4 cc per Kg for first 10 Kg, 2 cc per Kg for next 10 Kg and 1 cc per Kg for the next Kg of weight) calculated based on the patient's weight
- Ondansetron - Control Group: The control group received Dexamethasone (dose 0,15 mg/Kg) as standard antiemetic prophylaxis. Ondansetron (dose 0,05 mg/Kg) was used as a second prophylactic antiemetic.
  Ondansetron (Control): Ondansetron was used at a prophylactic dose (0,05 mg per Kg) based on patient's weight.
Period: Overall Study
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
Started | 150 (Enrolment phase: Recruiting of participants started December 11, 2013) | 150 (Enrolment phase: Recruitment of participants started December 11, 2013)
Randomized (10 participants were excluded as did not meet the eligibility criteria) | 144 | 146
Completed | 108 (n=108 completed study and immediate follow up n=36 participants were lost to follow up at 24 hr) | 109 (n=109 completed study and immediate follow up n=37 participants were lost to follow up at 24 hr)
Not Completed | 42 | 41
Not completed — Did not meet elegibility criteria | 6 | 4
Not completed — Lost to Follow-up | 36 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group | Total
Number analyzed (Participants) | 144 | 146 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 144 | 146 | 290
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: Months] | 55 [47 to 68] | 56 [47 to 67] | 55 [47 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 74 | 144
  Male | 74 | 72 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 46 | 42 | 88
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 37 | 75
  More than one race | 5 | 11 | 16
  Unknown or Not Reported | 55 | 56 | 111
Weight (Kg) [Mean (Standard Deviation); unit: Kilograms] | 19.9 (4.9) | 20.0 (5.6) | 20 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Vomiting Between 0 to 2 Hours
Description: In the Post Anesthetic Care Unit (PACU) the proper data (intraoperative and recovery period) was recorded at immediate postoperative period, at 2 hours after the procedure and prior to discharge.
  Parents were informed during the consent process that postoperative 24 hour follow up was going to be done over the phone by researcher.
Time Frame: 0 to 2 hr after the procedure (in PACU)
Measure: Count of Participants; unit: Participants
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
Number analyzed (Participants) | 144 | 146
Participants | 11 | 5

2. Secondary Outcome: Number of Participants Receiving Rescue Antiemetic Medications
Description: Parents were informed during the consent process that postoperative 24 hour follow up was going to be done over the phone by the researcher.
  The number of participants (parents / caregivers) who answered the call was recorded, and from those the number of patients who presented the secondary outcome.
Time Frame: 2 to 24 hr after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
Number analyzed (Participants) | 108 | 109
Participants | 15 | 9

3. Other Pre Specified Outcome: Number of Participants Having Delayed Home Discharge
Description: Data was recorder for number of patients with delays in discharge from PACU due to POV
Time Frame: Within 24 hours after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
Number analyzed (Participants) | 144 | 146
Participants | 2 | 0

4. Other Pre Specified Outcome: Blood Glucose Level
Description: Measuring the blood glucose level is important to ensure that administration of IV Dextrose at the dose to be used in our protocol, did not cause hyperglycemia in the participants. This measurement was done while patients were still under general anesthetic during the procedure.
Time Frame: Intraoperatively
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
Number analyzed (Participants) | 144 | 146
mmol/L | 6.3 [5.3 to 7.1] | 5.5 [4.8 to 6.0]

ADVERSE EVENTS:
Time Frame: Within 24 hours of administration of intervention (D5NS) vs Ondansetron.
Arm/Group | Dextrose (D5NS) - Intervention Group | Ondansetron - Control Group
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/146
Other Adverse Events (participants affected / at risk) | 0/144 | 0/146

LIMITATIONS AND CAVEATS:
No true placebo arm (unethical to withhold PONV prophylaxis) Inability to record or analyze the incidence of post-operative nausea This study was underpowered - size estimation Lack of a standardized anesthetic protocol minimized by randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No